CLINICAL TRIAL: NCT02681731
Title: Impact of Neuromonitoring During Cardiothoracic Procedures: A Retrospective Analysis
Brief Title: Impact of Neuromonitoring During Cardiac Procedures
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Delirium; Stroke; Acute Kidney Injury
MeSH Terms: conditions — Delirium; Stroke; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Through a series of sequential analyses, retrospective database exploration looking for linkages and associations between the use of processed electroencephalogram (EEG) and/or cerebral saturation monitoring and patient outcomes post-cardiothoracic surgery will be explored.

DETAILED DESCRIPTION:
The purpose of this study is to mine the Premier Healthcare Database to:

1. define the incidence of post-operative cognitive complications, acute kidney injury and stroke after specific cardiac surgical procedures (defined as: coronary artery bypass graft [CABG], Aortic Valve Replacement, Mitral valve repair, Mitral valve replacement, thoracic aortic operation, combined CABG and Valve replacement or repair ; and
2. Determine the incremental increase in the length of hospitalization and cost of hospitalization among cardiac surgical patients who suffer postoperative cognitive complications, acute kidney injury and stroke; and
3. Determine the effectiveness of intraoperative neuromonitoring with cerebral saturation and/or processed electroencephalogram (EEG) monitoring on the incidence of post-operative cognitive complications, acute kidney injury and stroke as a consequence of specific cardiac surgery procedures.

The Premier Healthcare Database is a privately owned database that represents approximately 1/5th of all United States hospitalizations annually. It includes all International Classification of Diseases-9th Revision (ICD-9) and International Classification of Diseases-Clinical Modification (ICD-9-CM) diagnosis and procedure codes recorded by the hospital, as well as a limited set of Current Procedural Terminology (CPT)-4 codes. Within the database, discharge-level data include information on patient and provider characteristics, diagnoses and procedures, hospital resource utilization, and charges/cost data for all entries, including pharmacy charges.

ELIGIBILITY:
Inclusion Criteria:

* All adult (age >=18 years) hospitalized patients who underwent major cardiac surgical procedure requiring cardiopulmonary bypass captured in the premier database from January 1, 2010 - December 31, 2014 (5 year period)

Exclusion Criteria:

* <18 years of age
* Cardiac procedures not requiring cardiopulmonary bypass

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult (age >=18 years) inpatients who underwent major cardiac surgical procedure requiring cardiopulmonary bypass captured in the Premier database from January 1, 2010 - December 31, 2014 (5 year period).
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Delirium: Incidence of post-operative cognitive complications identified by ICD-9 diagnosis code | 5 years
  Incidence of post-operative cognitive complications identified by International Classification of Disease (ICD-9) diagnosis code
Acute Kidney Injury: Incidence of acute kidney injury identified by ICD-9 diagnosis code | 5 years
  Incidence of acute kidney injury identified by ICD-9 diagnosis code
Stroke: Incidence of stroke identified by ICD-9 diagnosis code | 5 years
  Incidence of stroke identified by ICD-9 diagnosis code

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shaw, MB FRCA, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University School of Medicine, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
There is no individual participant data in this retrospective database study.